CLINICAL TRIAL: NCT00541645
Title: Transient Osteoporosis of Pregnancy: A Possible Peptide Mediator
Status: Suspended | Type: Observational
Sponsor: Hadassah Medical Organization (Other)
Other Study IDs: Lib001-HMO-CTIL
Record Dates: First submitted 2007-10-07; First posted 2007-10-10 (Estimated); Last update posted 2008-03-18 (Estimated); Status verified 2008-03

CONDITIONS: Transient Osteperosis

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Transient osteoporosis of pregnancy (TOoP) is uncommonly encountered in orthopedic and obstetric practice, with most reports consisting of single cases.

This rare condition consists of significant osteoporosis affecting the hips and spine, causing significant morbidity, and putting young female patients at risk for vertebral and femoral neck fractures.

The pathogenesis of transient osteoporosis of pregnancy is unknown, with various theories as to its etiology.

Recently, a number of reports have described elevated levels of PTHrP in patients with transient osteoporosis in pregnancy and of the postpartum period Our goal in this study is to assess the role of PTHrP in transient osteoporosis of pregnancy

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed consent

Ages: 18 Years to 45 Years | Sex: Female
Age Groups: Adult

CONTACTS AND LOCATIONS:
Overall Officials: Efrain Liebner, MD, Principal Investigator — Hadassah Medical Organization; Meir Liebergall, M.D, Study Chair — Hadassah Medical Organization; Tzvi Bar-Shavit, Ph.D, Study Director — The Hebrew University